CLINICAL TRIAL: NCT00132353
Title: Clinical Neurophysiology: Training and Normative Values
Brief Title: Training for Diagnosing Neurological Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050223; 05-N-0223
Record Dates: First submitted 2005-08-18; First posted 2005-08-19 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Musculoskeletal Physiology
Keywords: Magnetic Stimulation; Single Fiber EMG; Ultrasonography; Autonomic Testing; Near-nerve recording

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (2):
- Healthy volunteers: For normative data
- Patients with neurological disorders: For teaching fellows electrodiagnostic techniques

SUMMARY:
This training protocol has two objectives: 1) to train NINDS fellows in specialized techniques for diagnosing neurological disorders, and 2) to gather data from healthy volunteers and from patients with various disorders needed for tests to diagnose disorders of nerve, muscle, and the areas of the brain controlling movement.

Healthy volunteers and patients with neurological disorders of nerve and muscle who require specialized diagnostic testing may be eligible for this study. Candidates must be 18 years of age or older. They are screened with a medical history and neurological examination.

Immediately after screening, participants undergo one or two of the following tests:

* Transcranial magnetic stimulation: This procedure maps brain function. A wire coil is held on the scalp, and a brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. During the stimulation, the subject may be asked to tense certain muscles slightly or perform other simple actions. The stimulation may cause a twitch in muscles of the face, arm, or leg, and the subject may hear a click and feel a pulling sensation on the skin under the coil. During the stimulation, electrical activity of muscles is recorded with a computer, using electrodes (small metal disks) attached to the skin with tape.
* Electromyography (EMG): This test measures the electrical activity of muscles and is used to diagnose problems with the nerves or muscles. For surface EMG, electrodes are filed with a conductive gel and taped to the skin. Needle EMG involves inserting a needle into a muscle to record the electrical activity. Single fiber EMG uses specialized needles that allow recording from single muscle fibers. The needle is inserted into a muscle and the subject is asked to tense that muscle slightly.
* Nerve conduction study: This test measures the speed with which nerves conduct electrical impulses and the strength of the connection between the nerve and the muscle. It is done by taping wires on the skin to record the impulses and placing a probe on the skin to deliver a small electrical stimulus.
* Near-nerve recording: This test is a nerve conduction study that is used to measure responses from very small nerves. It uses a needle placed under the skin to record the nerve response.
* Quantitative sensory testing: This test measures how well the subject feels vibration and cold. A probe that can vibrate or cool down is attached to the subject's finger or foot. The subject presses a button when he or she feels the stimulus. A computer adjusts the intensity of the stimulus to find the lowest level the subject can feel.
* Nerve ultrasound: This test uses sound waves to examine the nerves. Warm gel is applied to the skin and a probe is held on the skin surface.

DETAILED DESCRIPTION:
Objective: This is a training protocol. The goal of this protocol is to train fellows in advanced physiological techniques used for diagnosing neurological disorders. A secondary objective of the protocol is to gather normative data for diagnostic neurophysiologic tests.

Study population: Patients and healthy adult volunteers may be studied under this protocol. Patients must have a clinical indication for the diagnostic test. Most patients will be enrolled in a primary NIH protocol, and this protocol will serve as a secondary protocol. Occasionally, patients will be enrolled in this protocol as a primary protocol when they are referred from hospitals that participate in the NINDS fellowship training program. Healthy adults will be studied by fellows-in-training to practice a new testing procedure or to provide normative data when required by changes in instrumentation or laboratory technique.

Design: Testing will be performed during an outpatient clinic visit. One or two of the following procedures may be performed as clinically indicated: single fiber EMG, macro-EMG, near-nerve recording, single-pulse transcranial or peripheral nerve magnetic stimulation, quantitative sensory testing, nerve conduction studies, electromyography, nerve ultrasonography, or autonomic testing.

Outcome measures: This is a training protocol. No research will be carried out under this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA FOR PATIENTS:

Adult patients, over age 18 years old, with a clinical indication for the diagnostic procedures will be enrolled

* Suspected disorders of neuromuscular transmission, such as myasthenia gravis or
* Suspected Central demyelinating disorders such as multiple sclerosis or
* Suspected Myelopathy or
* Suspected motor neuron disease or
* Suspected Movement disorders that impair intracortical processes or
* Suspected neuropathy or myopathy or
* Suspected autonomic dysfunction

INCLUSION CRITERIA FOR HEALTHY VOLUNTEERS:

Healthy adults, aged 18 years or older, willing to participate

EXCLUSION CRITERIA FOR PATIENTS:

* Patients with implanted devices, such as pacemakers, or metal in the cranium (excluding dental work) will be excluded from magnetic stimulation studies.
* Children under age 18 will be excluded, since the goal of this protocol is to provide training experience.
* Subjects who are unable to provide informed consent
* Persons undergoing the autonomic testing will be asked to refrain from smoking, caffeine, alcohol and vigorous exercise 24 hours before the study. Several medications should not be taken 48 hours prior to the study; these include tricyclic antidepressants, antihistamines, cough and cold medications, anti-Parkinson medication, muscle relaxants, anti-psychosis medications, opioid drugs, and blood pressure medications. No one is to stop their prescribed medication without discussion with their primary care physician though the ability to complete all of the autonomic testing may be affected.

EXCLUSION CRITERIA FOR HEALTHY VOLUNTEERS:

* Medical conditions that require medications that affect the physiological measures being tested
* History of stroke, peripheral neuropathy or spine surgery
* Implanted devices or metal in the cranium (except dental work) if undergoing magnetic stimulation
* Persons undergoing the autonomic testing will be asked to refrain from smoking, caffeine, alcohol and vigorous exercise 24 hours before the study. Several medications should not be taken 48 hours prior to the study; these include tricyclic antidepressants, antihistamines, cough and cold medications, anti-Parkinson's medication, muscle relaxants, anti-psychosis medications, opioid drugs, and blood pressure medications. No one is to stop their prescribed medication without discussion with their primary care physician and you may be excluded from the study.
* NIH employees and staff may participate, except if they are EMG Section, OCD, NINDS employees.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal volunteers and individuals with neurological disorders amenable to diagnosis through electrodiagnostic techniques.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2005-11-04 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya J Lehky, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2005-N-0223.html